CLINICAL TRIAL: NCT05407324
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating Safety and Efficacy of CORT113176 (Dazucorilant) in Patients With Amyotrophic Lateral Sclerosis (DAZALS)
Brief Title: Dazucorilant in Patients With Amyotrophic Lateral Sclerosis
Acronym: DAZALS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CORT113176-652; 2021-005611-31 (EudraCT Number)
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS, Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — CORT113176

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: CORT113176 (Dazucorilant) 300 mg (Experimental): 300 mg of dazucorilant will be administered once daily.
  Interventions: Drug: Dazucorilant 300 mg
- Part 1: CORT113176 (Dazucorilant) 150 mg (Experimental): 150 mg of dazucorilant will be administered once daily.
  Interventions: Drug: Dazucorilant 150 mg; Other: Placebo
- Part 1: Placebo (matched to study drug) (Placebo Comparator): Placebo will be administered once daily.
  Interventions: Other: Placebo
- Part 2: CORT113176 (Dazucorilant) 75 - 300 mg Dose-titration (Experimental): 75 mg of dazucorilant will be administered once daily for 1 week, and increased weekly in 75 mg increments up to 300 mg once daily.
  Interventions: Drug: Dazucorilant

INTERVENTIONS:
Drug: Dazucorilant 300 mg — 300 mg of dazucorilant will be administered once daily in 4 capsules of 75 mg dazucorilant/capsule.
  Other Names: CORT113176
  Arms: Part 1: CORT113176 (Dazucorilant) 300 mg
Drug: Dazucorilant 150 mg — Dazucorilant and placebo will be administered once daily in 4 capsules, 2 capsules with 75 mg dazucorilant/capsule, and 2 capsules of placebo equivalent.
  Other Names: CORT113176
  Arms: Part 1: CORT113176 (Dazucorilant) 150 mg
Other: Placebo — Placebo will be administered once daily in capsules of placebo equivalent.
  Arms: Part 1: CORT113176 (Dazucorilant) 150 mg; Part 1: Placebo (matched to study drug)
Drug: Dazucorilant — Dazucorilant will be administered once daily in 75-mg capsules.
  Other Names: CORT113176
  Arms: Part 2: CORT113176 (Dazucorilant) 75 - 300 mg Dose-titration

SUMMARY:
The purpose of this 2-part study is to assess the safety and efficacy of CORT113176 (dazucorilant) in patients with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
In Part 1, eligible ALS patients will be randomized to one of three treatment arms (1:1:1) across North America and Europe for a 24-week double-blind treatment period. Patients who complete participation (i.e., completed all visits) in the double-blind treatment period will be eligible for participation in a 132-week open-label extension (OLE) study. A daily dose of 300 mg dazucorilant will be used in the 132-week OLE period. Patients who complete the double-blind treatment period and who do not enter the OLE will enter the 132-week follow-up period.

In Part 2, eligible ALS patients will receive open-label treatment to evaluate dose titration and tolerability of dazucorilant. The dose titration will begin with an initial 75 mg once daily dose, and the dose will be titrated up as tolerated in 75 mg increments until the 300 mg once daily target dose is reached and maintained for 3 weeks. Patients who complete participation in the dose-titration treatment period will be eligible to continue treatment with dazucorilant 300 mg once daily in a 52-week open-label extension portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years of age with Sporadic or familial ALS. In Part 1, patients must have a risk of ALS progression characterized by a European Network for the Cure of ALS (ENCALS) risk profile score ≥ -6 and ≤ -3. In Part 2 patients must have a risk of ALS progression characterized by an ENCALS risk profile score ≥ -7 and ≤ -3.
* If taking riluzole, edaravone, and/or sodium phenylbutyrate and taurursodiol, must be on a stable dose prior to Screening. Sodium phenylbutyrate and taurursodiol are not permitted for patients enrolled in Part 2 of the study.
* Part 2 only: Patients with a pathogenic mutation in superoxide dismutase 1 gene (SOD1) must not be receiving treatment with tofersen or eligible for treatment with tofersen if available. Patients who have received prior treatment with tofersen and discontinued due to safety and/or efficacy reasons prior to Screening are eligible.
* Part 2 only: Use of ultra high-dose methylcobalamin for the treatment of ALS is permitted provided the patient has been on a stable dose for ≥11 weeks prior to the Day 1 visit.

Exclusion Criteria:

* History of a clinically significant non-ALS neurologic disorder
* Inability to swallow capsules.
* Blood platelet count <150,000/mm^3.
* Renal impairment indicated by Estimated Glomerular Filtration Rate (eGFR) ≤30 mL/min/1.73 m^2. Part 2 only: Patients with a recent history of acute kidney injury should have returned to their baseline renal function prior to enrollment.
* Human immunodeficiency virus (HIV) or current chronic/active infection with hepatitis C virus or hepatitis B virus. Part 2 only: Known history of HIV or chronic/active infection with hepatitis C or hepatitis B virus; testing does not need to be performed if infection status is unknown.
* Women who are pregnant, planning to become pregnant, or are breastfeeding.
* Use of non-invasive ventilation (NIV) or mechanical ventilation via tracheostomy, or on any form of oxygen supplementation.
* Current or anticipated need of a diaphragm pacing system (DPS).
* Currently using glucocorticoids or have a history of regular systemic glucocorticoid use within the last 12 months.
* Previous exposure or treatment with glucocorticoid receptor modulators or antagonists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 24 in the ALS Functional Rating Scale-Revised (ALSFRS-R) total score. | Baseline to Week 24
  This outcome measure is assessed in study Part 1.
Incidence of Adverse Events (AEs), Serious Adverse Events (SAEs), treatment-related AEs, AEs by severity, and deaths due to AEs | Baseline to Week 24
  This outcome measure is assessed in study Part 1.
Incidence of treatment-emergent AEs and SAEs | Baseline up to Week 12
  This outcome measure is assessed in study Part 2.
Incidence of treatment-emergent AEs leading to dose interruptions, dose reductions, and/or discontinuations of study drug | Baseline up to Week 12
  This outcome measure is assessed in study Part 2.

SECONDARY OUTCOMES:
Change from Baseline to Week 24 in muscle strength (assessed using hand-held dynamometer) | Baseline to Week 24
  This outcome measure is assessed in study Part 1.
Change from Baseline to Week 24 in Percent Slow Vital Capacity | Baseline to Week 24
  This outcome measure is assessed in study Part 1.
Change from Baseline to Week 24 in EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) | Baseline to Week 24
  This outcome measure is assessed in study Part 1.
Time to Death | From randomization date to the date of death from any cause up to 156 weeks
  This outcome measure is assessed in study Part 1.

CONTACTS AND LOCATIONS:
Overall Officials: Corcept Therapeutics Incorporated, Study Director — Corcept Therapeutics Incorporated
Locations (35):
- United States (4):
  - 062, Phoenix, Arizona
  - 278, San Francisco, California
  - 287, Neptune City, New Jersey
  - 353, New York, New York
- 108, Leuven, Belgium
- Canada (2):
  - 425, Hamilton, Ontario
  - 273, Montreal, Quebec
- France (8):
  - 422, Bron
  - 258, Lille
  - 257, Limoges
  - 261, Marseille
  - 423, Montpellier
  - 259, Nice
  - 262, Paris
  - 256, Tours
- Germany (8):
  - 255, Berlin
  - 270, Bonn
  - 268, Dresden
  - 260, Hanover
  - 265, Jena
  - 386, München
  - 267, Rostock
  - 269, Ulm
- 253, Dublin, Ireland
- 264, Utrecht, Netherlands
- Poland (4):
  - 283, Bydgoszcz
  - 385, Krakow
  - 254, Warsaw
  - 274, Warsaw
- Spain (5):
  - 302, Barcelona
  - 115, Barcelona
  - 303, Madrid
  - 282, Málaga
  - 194, Valencia
- 263, Stoke-on-Trent, United Kingdom

IPD SHARING:
Plan to Share IPD: No